CLINICAL TRIAL: NCT06410885
Title: Assessment of Flow in Cerebrospinal Fluid Shunts With a Wireless Thermal Anisotropy Measurement Device in Asymptomatic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhaeos, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-03
Record Dates: First submitted 2024-05-03; First posted 2024-05-13 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Observational, part 1 (blinded) (Experimental)
  Interventions: Device: Thermal Anisotropy Measurement Device
- Diagnostic, part 2 (unblinded) (Experimental)
  Interventions: Device: Thermal Anisotropy Measurement Device

INTERVENTIONS:
Device: Thermal Anisotropy Measurement Device — The study device is a non-invasive sensor that is placed on the study subject's skin overlying an existing implanted CSF shunt. It uses an integrated thermal actuator and temperature sensors to assess shunt flow.

SUMMARY:
This study evaluates the performance of the study device, FlowSense®, a sensor for non-invasively assessing cerebrospinal fluid (CSF) shunt flow. Subjects with an existing implanted ventricular CSF shunt will be evaluated with the study device in an outpatient setting to determine the negative predictive value (NPV; Part 1, blinded) and explore changes in surveillance imaging, health resource utilization, and visit duration during routine follow-up visits (Part 2, unblinded).

ELIGIBILITY:
Inclusion criteria

1. Existing ventricular cerebrospinal fluid shunt
2. Age ≥ 2 years old
3. Region of intact skin overlying an unambiguously identifiable palpable chronically indwelling ventricular shunt that crosses the clavicle; region of skin is appropriate in size for application of the study device
4. Capable of providing informed consent or have a legal guardian, health care agent, or surrogate decision-maker able to provide informed consent
5. Standard of care outpatient visit with neurosurgeon assessment of having "no clinical concern for shunt malfunction"

Exclusion criteria

1. Subject not scheduled to receive outpatient standard of care imaging (CT, MRI, X-ray shunt series) as part of the clinic visit
2. Presence of more than one distal shunt catheter in the study device measurement region
3. Presence of an interfering open wound or edema in the study device measurement region
4. Subject-reported history of adverse skin reactions to silicone adhesives
5. Participation in the study will interfere with, or be detrimental to, the administration of optimal health care to the subject
6. Subject not available for seven-day follow-up

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Study device negative predictive value (NPV) | Up to 7 days
  The study device will produce either "flow confirmed" or "flow not confirmed" data in a blinded fashion. Ground truth will be established based on 7-day follow-up an intraoperative observations for any surgery performed per the standard of care.

SECONDARY OUTCOMES:
Study device sensitivity, specificity, diagnostic accuracy, and positive predictive value (PPV) | Up to 7 days
  The study device will produce either "flow confirmed" or "flow not confirmed" data in a blinded fashion. Ground truth will be established based on 7-day follow-up an intraoperative observations for any surgery performed per the standard of care.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Benioff Children's Hospital, San Francisco, California, United States